CLINICAL TRIAL: NCT01258439
Title: Post-prandial Lipid Effects of Raltegravir (RAL) vs Ritonavir-boosted Darunavir (DRV-r) in Anti-retroviral Therapy (ART)-Naive Adults or Adults Recommencing ART.
Brief Title: Post-prandial Lipid Effects of Raltegravir (RAL) vs Ritonavir -Boosted Darunavir (DRV-r) in Anti-retroviral Therapy (ART)- Naive Adults or Adults Recommencing ART.
Acronym: ROaR+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Andrew Carr, Head, Clinical Research Program, St Vincent's Hospital, Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROaR+
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: HIV; Cardiovascular Disease
Keywords: HIV; cardiovascular disease; post prandial lipids; ritonavir; darunavir; raltegravir; arterial stiffness; tonometry
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Darunavir; Ritonavir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.Raltegravir plus truvada (Active Comparator): Raltegravir 400mg twice daily plus truvada 300mg/200mg once daily for 24 weeks
  Interventions: Drug: Darunavir, ritonavir, tenofovir/emtricitabine (Truvada)
- 2. ritonavir boosted darunavir plus truvada (Active Comparator): Darunavir 800mg with ritonavir 100mg plus truvada 300mg/200mg once daily for 24 weeks
  Interventions: Drug: raltegravir plus truvada

INTERVENTIONS:
Drug: raltegravir plus truvada — raltegravir 400 mg tablet with truvada 300/200 mg tablet for 24 weeks
  Other Names: tenofovir disoproxil fumarate; Isentress
  Arms: 2. ritonavir boosted darunavir plus truvada
Drug: Darunavir, ritonavir, tenofovir/emtricitabine (Truvada) — Darunavir two 400mg tablets with one ritonavir 100mg capsule once daily plus Tenofovir/emtricitabine (Truvada) one 300mg/200mg tablet once daily with food for 24 weeks
  Other Names: Prezista; Norvir; Tenofovir/emtricitabine
  Arms: 1.Raltegravir plus truvada

SUMMARY:
This is a research study into the effects of three drugs used to treat HIV infection. Some drugs used to treat HIV have been associated with changes in blood fats such as cholesterol that could be harmful over the long-term, because these blood fat changes have been associated with a small, increased risk of heart disease and stroke in some studies of adults with HIV. Now that HIV can be controlled for long periods in most patients, and because heart disease is one of the biggest causes of illness and death in the general population, it is important to develop new HIV treatments that control HIV effectively but do not cause abnormal blood fats.

Hypothesis: That Raltegravir will result in less post-prandial lipid disturbances than ritonavir-boosted darunavir.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, informed consent
* Age >18 years
* HIV infection documented by HIV antibody test and Western Blot prior to study entry
* No previous ART OR no ART for 6 months prior to randomisation
* CD4+ count of <500 cells/mm or viral load >10,000 copies/ml within 60 days prior to randomisation
* No genotypic resistance to Raltegravir, Tenofovir/emtricitabine, Darunavir, Ritonavir
* Body mass index less than 30kg/m2

Exclusion Criteria:

* Primary HIV infection within the last 6 months
* Active infection or opportunistic illness within the previous 30 days
* Use of any medication contra-indicated with ritonavir-boosted darunavir or raltegravir
* Use of lipid-lowering therapy
* Diabetes mellitus (fasting glucose >7.0mml/l or a prior diagnosis of diabetes)
* Use of oral prednisolone > 7.5mg daily or equivalent
* pregnancy or Breast feeding
* proven hypersensitivity to one or more components of the study meal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To compare the effects of ritonavir plus darunavir daily to raltegravir twice daily on post prandial lipid responses over 24 weeks | 24 weeks
  Fasting samples will be taken for total cholesterol, LDL and HDL cholesterol, and triglycerides. Repeat lipid samples will be collected before a high fat meal is consumed. After the meal is completed , blood will be collected at 1, 2, 3, and 4 hours at baseline, week 4 and week 24 visits.

SECONDARY OUTCOMES:
safety | 24 weeks
  Safety parameters will be assessed by measurement of urea and electrolytes, LFTs, urine protein to creatinine ratio
Other metabolic parameters | 24 weeks
  Fasting metabolic parameters will be assessed. Study staff and participants will be blinded to the results fo these tests until completion of the study or parameters become sginificantly abnormal
Arterial stiffness | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Carr, Professor, Principal Investigator — St Vincent's Hospital - Sydney, Australia
Locations (2):
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - St Vincent Hospital, Clinical Research Program, Sydney, New South Wales